CLINICAL TRIAL: NCT07104149
Title: Neoadjuvant Chemotherapy Plus Cadonilimab for Locally Advanced Cervical Cancer : a Multicentre, Single Arm, Phase 2 Trial
Brief Title: Neoadjuvant Chemotherapy Plus Cadonilimab for Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Second Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Ya, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-MA-0101
Record Dates: First submitted 2025-03-31; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Female, Age ≥ 18 Years Old; No Previous Systemic Treatment for the Current Disease, Including Surgery, Antitumor Radiochemotherapy/Immunotherapy; ECOG Score of 0-1; Histologically Confirmed Cervical Cancer, FIGO Stage IB3, IIA2, IIB, IIIC, and Assessed by the Researcher as Resectable Lesion; Sufficient Organ Function; The Result of the Urine or Serum Pregnancy Test for the Subject is Negative; Subjects Should Take Contraceptive Measures; Locally Advanced Cervical Cancer; Expected Survival Time >6 Months
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy plus cadonilimab for locally advanced cervical cancer (Experimental): Cadonilimab 10mg/kg, ivgtt., D1, q3w with Cisplatin ( 75mg/ m2, ivgtt., D2, q3w) for a total of 2-4 cycles before radical surgical treatment.
  Interventions: Drug: Cadonilimab combined with cisplatin

INTERVENTIONS:
Drug: Cadonilimab combined with cisplatin — Neoadjuvant chemotherapy plus cadonilimab for locally advanced cervical cancer

SUMMARY:
Main Purpose of this study is to determine the efficacy and safety of Cadonilimab combined with chemotherapy (cisplatin) for locally advanced cervical cancer.

This is an multicentre, single Arm, Phase 2 Trial study of Cadonilimab with Cisplatin in the treatment of locally advanced cervical cancer. 29 eligible patients will receive Cadonilimab（10mg/kg, iv., D1, q3w）with Cisplatin ( 75mg/ m2, iv., D2， q3w) for a total of 2-4 cycles before radical surgical treatment.

DETAILED DESCRIPTION:
Detailed Description:

Study Title : Neoadjuvant Chemotherapy Plus Cadonilimab for Locally Advanced Cervical Cancer : a Multicentre, Single Arm, Phase 2，prospective Trial Main Study Objectives : Determine the efficacy and safety of Cadonilimab combined with chemotherapy (cisplatin) for locally advanced cervical cancer.

Secondary Objective: Explore the correlations between the expression of PD-L1 , Tumor Mutational Burden（TMB） levels, immune cell subsets, tumor microenvironment and therapeutic efficacy

Study Endpoints :

Primary Endpoint :Pathological complete response rate (pCR) and Radiological response rate (RS) Secondary Endpoints :Safety (Incidence and severity of adverse events (AE) caused by drug treatment and perioperative complications, clinically significant abnormal laboratory test results;Clinical downstaging rate (downstaging of T and/or N); Major pathological response rate (MPR);Disease-free survival (DFS); Objective response rate (ORR) ,Disease control rate (DCR), progression-free survival (PFS), and 5-year overall survival rate (OS) based on RECIST v1.1 and mRECIST evaluation.

Target Population : Patients with histologically confirmed cervical cancer , stage IB3, IIA2, IIB, and IIIC according to FIGO , and the lesion was resectable .

Study Drug and Administration . 29 eligible patients will receive Cadonilimab（10mg/kg, ivgtt., D1, q3w）with Cisplatin ( 75mg/ m2, ivgtt., D2，q3w) for a total of 2-4 cycles before radical surgical treatment. Dose adjustments are not allowed during the treatment ,Treatment may be delayed for a maximum of 12 weeks from the previous treatment.

Imaging examinations were conducted to evaluate the efficacy of neoadjuvant therapy and the possibility of radical resection. Radical surgery for cervical cancer was then performed. The study investigators would determine whether adjuvant therapy was necessary and select an appropriate treatment plan (the first treatment was initiated 6 weeks ± 2 weeks after surgery and could not exceed 3 months). Imaging evaluations were conducted every three months after surgery until disease recurrence. Survival follow-up was performed every three months after disease recurrence. Safety visit: From the first administration of medication to 60 days after the last administration or the initiation of new anti-tumor treatment.

ELIGIBILITY:
Histologically confirmed cervical carcinoma, FIGO stage IB3, IIA2, IIB, IIIC1, and assessed as resectable by the researcher。

Inclusion Criteria:

* Female, age ≥18 years;
* Histologically confirmed cervical cancer, FIGO stage IB3, IIA2, IIB, IIIC, and assessed by the researcher as resectable;
* No previous systemic treatment for the current disease, including surgical treatment, antitumor chemoradiotherapy/immunotherapy, etc.;
* Patients who agree to undergo radical surgical treatment and are judged by the surgeon to have no surgical contraindications;
* ECOG score of 0-1;
* Expected survival time >6 months;
* Sufficient organ function, the subject must meet the following laboratory indicators:

Neutrophil absolute count (ANC) ≥1.5x10^9/L ; Platelets ≥100x10^9/L ;Hemoglobin >9g/dL ; Total bilirubin ≤1.5× upper limit of normal (ULN); Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN; Serum creatinine ≤1.5×ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 ml/min; international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; Normal thyroid function; Myocardial enzymes within the normal range

Exclusion Criteria:

* Diagnosis of other malignancies within 5 years prior to the first dose (excluding adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone radical resection).
* Current participation in an interventional clinical study or receipt of other investigational drugs or devices within 4 weeks prior to the first dose.
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or drugs targeting other stimulatory or co-inhibitory T-cell receptors .
* Systemic treatment with Chinese herbal medicines with antitumor indications or immunomodulatory agents (e.g., thymosin, interferon, interleukin, excluding local use for pleural effusion control) within 2 weeks prior to the first dose.
* Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapies (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal/pituitary insufficiency) are not considered systemic treatment.
* Systemic glucocorticoid therapy (excluding nasal sprays, inhalations, or other local routes) or any immunosuppressive therapy within 7 days prior to the first dose.
* History of allogeneic organ transplantation (excluding corneal transplants) or allogeneic hematopoietic stem cell transplantation.
* Known hypersensitivity to any study drug.
* Presence of multiple factors affecting cisplatin use (e.g., platinum allergy).
* Inadequate recovery from prior intervention-related toxicity or complications (i.e., >Grade 1 or not returned to baseline, excluding fatigue or alopecia).
* Known history of Human Immunodeficiency Virus（ HIV） infection .
* Untreated active hepatitis B （HBV）(defined as HBsAg-positive with HBV-DNA exceeding the upper limit of normal at the study site).
* Active hepatitisC (HCV) infection (HCV antibody-positive with HCV-RNA above the lower detection limit).
* Administration of live vaccines within 30 days prior to the first dose (Cycle 1, Day 1).
* Pregnant or lactating women.
* Severe or uncontrolled systemic diseases, including:Symptomatic resting Electrocardiograph abnormalities (e.g., complete left bundle branch block, ≥Grade II heart block, ventricular arrhythmia, atrial fibrillation).Unstable angina, congestive heart failure, or chronic heart failure ≥NYHA class II.Arterial thromboembolism, ischemia, myocardial infarction, unstable angina, stroke, or transient ischemic attack within 6 months prior to enrollment.Poorly controlled hypertension (systolic >140 mmHg, diastolic >90 mmHg).History of non-infectious pneumonitis requiring glucocorticoids within 1 year or current active interstitial lung disease.
* Active tuberculosis.
* Active or uncontrolled infection requiring systemic therapy.
* Clinically active diverticulitis, abdominal abscess, or gastrointestinal obstruction.
* Liver diseases (e.g., cirrhosis, decompensated liver disease, acute/chronic active hepatitis).
* Poorly controlled diabetes (fasting blood glucose >10 mmol/L).
* Urine protein ≥++ on urinalysis with 24-hour urine protein >1.0 g.
* Psychiatric disorders impairing compliance.
* Any condition (e.g., medical history, abnormal lab/test results, concurrent treatments) that may interfere with study outcomes, participation, or pose risks, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | From enrollment to 5 years after the end of treatment
  The proportion of subjects with no residual viable tumor cells and negative lymph nodes among all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Xie Ya, Study Chair — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No